CLINICAL TRIAL: NCT06207162
Title: Longitudinal Neural Fingerprinting of Opioid-use Trajectories
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2000036564; 1R21DA058415-01A1 (NIH)
Record Dates: First submitted 2023-12-19; First posted 2024-01-16 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Opioid Use Disorder
Keywords: Medication for Opioid Use Disorder (MOUD)
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- neural fingerprinting of MOUD (Experimental): Study participants will have one in-person screening (2 hours), 6 in-person visits for fMRI scans conducted biweekly (4 hours), and will be computationally assessed 12 times, once per week for 12 weeks. After participation in the main study, participants will be asked to complete a 15-minute follow up every month for an additional three months
  Interventions: Diagnostic Test: fMRI

INTERVENTIONS:
Diagnostic Test: fMRI — Participants will be performing tasks while undergoing fMRI. Tasks include Stroop task, Emotion-regulation task and an Ambiguity reward task. There will also be a Resting state: Participants are not presented with any specific stimulus.

SUMMARY:
This project aims to collect a densely sampled neuroimaging dataset among individuals receiving medications for opioid use disorder (MOUD). MOUD is multiphasic, comprised of medication induction, stabilization, ongoing treatment, and eventual dis-continuation phases. However, with a few small exceptions, existing neuroimaging efforts are almost exclusively single time-point assessments which, by definition, fail to capture these clinically relevant transitions and thus also do not capture individual risk and resilience trajectories. The investigators innovation, the characterization of neurocomputational trajectories during clinically relevant phases of MOUD treatment, will provide unprecedented mechanistic insight into the neurobiological basis of recovery. Once characterized, such trajectories may be used in the identification of specific therapeutic windows for additional intervention (e.g., times of increased neural plasticity) and in the design of novel tailored interventions based on known brain mechanisms (e.g., behavioral therapy, neurostimulation, neurofeedback).

DETAILED DESCRIPTION:
MOUD individuals between the ages of 18 and 50 who recently enrolled in methadone treatment at APT Foundation clinics in the greater New Haven area. Investigators will aim to recruit individuals as early as possible in treatment, but individuals may be within the first 6 months of treatment at the time of screening, as this may be necessary to ensure that they are on a stable dose of methadone.

AIM 1 - Longitudinal neural fingerprinting of MOUD to repeatedly characterize neural trajectories of individuals in early methadone treatment.

AIM 2 - Complementary, longitudinal computational phenotyping of MOUD to repeatedly characterize behavioral, computational trajectories of individuals in early methadone treatment.

After participation in the main study, participants will be asked to complete a 15-minute follow up every month for an additional three months.

ELIGIBILITY:
Inclusion Criteria:

* within the first 6 months of methadone treatment for OUD and on a stable dose of methadone
* eligibility for MRI scanning
* willing to commit to longitudinal study visits

Exclusion Criteria:

* current psychosis, mania, or suicidal ideation with intent, as assessed during screening with the SCID-5
* current co-occurring severe substance-use disorders (excluding nicotine and opioids), as assessed during screening with the SCID-5
* current intoxication or acute withdrawal at time of study visit sufficient to prevent participation based on: behavioral observation, breathalyzer, and SOWS assessment (these individuals will be allowed to enroll at a later date once stable)
* severe cognitive impairment (determined through consent process conducted by trained clinical research staff and during consent quiz or as indicated by a PROMIS Cognitive Function t-score <30 (i.e., score indicating severe impairment)
* Past or present history of intellectual disability or developmental disorder
* Neurological disease (including seizures or epilepsy) as assessed by self-report and by consulting clinic records
* Head trauma with loss of consciousness of more than 30 minutes
* Organ dysfunction or any unstable or untreated medical conditions that may alter cerebral function or interfere with study participation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in Relationship between functional connectivity within canonical neural networks and within the 'opioid abstinence network' and opioid use | up to 12 weeks
  Relationship between functional connectivity within canonical neural networks and within the 'opioid abstinence network' and opioid use over 6 biweekly sessions. Functional connectivity is computed as the Pearson's correlation between two brain regions, or 'nodes'. This will be done in a pairwise manner to obtain connectivity values for all possible node pairs in the Shen atlas, a 268-node atlas covering the cortex, subcortex and cerebellum. Correlation coefficients are transformed to Z-scores using Fisher's r-to-z transformation. Connectivity within a given network is defined as the mean of the Z values for all of the edges (connection between two node pairs) within the network.

SECONDARY OUTCOMES:
Change in Presence or absence of opioid use | up to 12 weeks
  Relationship between performance on the risk and ambiguity task and opioid use over 12 weekly sessions. Parameters are computed from the participant's choice data during task performance at each weekly time point. The primary task parameter is α. This is a participant-specific known-risk tolerance parameter.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Yip, PhD, MSc, Principal Investigator — Yale University
Locations (1):
- MRRC at The Anlyan Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will submit and share data with OpenNeuro. This will include de-identified demographic data, neuropsychological assessment data, clinical assessment data, and fMRI data (raw).
Time Frame: All data will be deposited to OpenNeuro starting 24 months after data collection begins and will be deposited every six months thereafter. OpenNeuro policy states that any data uploaded to their repository becomes publicly available under a Creative Commons CC0 license after a 36-month period beginning from first successful version of the dataset.
Access Criteria: OpenNeuro policy states that any data uploaded to their repository becomes publicly available under a Creative Commons (CC) license after a 36-month period beginning from first successful version of the dataset. Users create an account with OpenNeuro account in order to download BIDS formatted files and any associated metadata.